CLINICAL TRIAL: NCT07098208
Title: The Effect of Meditation on Exam Anxiety of Nursing Students
Brief Title: The Effect of Twin Heart Meditation on Exam Anxiety of Nursing Students
Acronym: exam anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Pouran Varvani Farahani, PhD in Pediatric Nursing, Department of Nursing, Faculty of Health Science, Cyprus International University,, Cyprus International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PVF2025CAM002
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Exam Anxiety; Meditation
Keywords: Nursing Students; Complementary Therapies; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants in this clinical trial are randomly assigned to one of two groups: an experimental group receiving Twin Heart Meditation and a control group receiving standard academic care. Both groups are observed in parallel throughout the study duration.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double-Blind (Investigator, Outcomes Assessor):
  To minimize bias, a double-blind approach is employed. The data are collected by the researcher, who remains unaware of group assignments, and the statistician performing the analysis is also blinded to the allocation. The data are analyzed as anonymous variables (x₁ and x₂) to preserve objectivity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twin Heart Meditation (Experimental): Behavioral: Twin Heart Meditation Participants in this group receive the Twin Heart Meditation intervention, a guided meditative technique based on the principles of loving-kindness and spiritual energy. The intervention is designed to reduce exam-related anxiety by promoting inner peace and emotional regulation.
  Interventions: Behavioral: Twin Heart Meditation
- Routine Academic Preparation (No Intervention): Participants in this group continue with their usual academic preparation and receive no additional interventions.

INTERVENTIONS:
Behavioral: Twin Heart Meditation — Participants in this group receive the Twin Heart Meditation intervention, a guided meditative technique based on the principles of loving-kindness and spiritual energy. The intervention is designed to reduce exam-related anxiety by promoting inner peace and emotional regulation. The meditation protocol follows the steps conceptualized by Master Choa Kok Sui and includes the following components:
  * Physical warm-up exercises
  * Activation of the heart chakra
  * Activation of the crown chakra
  * Blessing the Earth with loving-kindness
  * Silent meditation using the phrase "Amen"
  * Expression of gratitude
  * Closing exercises
  Participants practice the meditation in three guided sessions over one week, each lasting 30 minutes, under the supervision of a trained instructor. Sessions are conducted in a quiet room with audio guidance and follow-up support.
  Arms: Twin Heart Meditation

SUMMARY:
This randomized clinical trial aimed to evaluate the effectiveness of Twin Heart Meditation in reducing exam anxiety among undergraduate nursing students. The study focused on whether regular practice of this meditation technique could significantly reduce state anxiety before examinations. The main research questions were:

Does Twin Heart Meditation reduce exam-related anxiety among nursing students? Can this complementary and non-invasive method be considered a viable approach for managing academic stress? Participants were randomly assigned to either the intervention group, which practiced Twin Heart Meditation, or the control group, which followed routine academic activities. Pre- and post-intervention anxiety levels were measured using the State-Trait Anxiety Inventory (STAI).

DETAILED DESCRIPTION:
Study Title:

The Effect of Twin Heart Meditation on Exam Anxiety of Nursing Students

Study Purpose:

The aim of this study was to investigate the efficacy of Twin Heart Meditation a mind-body relaxation technique rooted in complementary and alternative medicine in reducing exam anxiety among undergraduate nursing students. The intervention was designed in accordance with holistic nursing principles and implemented in a controlled, double-blind randomized trial setting.Sample Size Determination:

The statistical population of this study included seventh-semester nursing students enrolled in the English-language program at Near East University. Out of 120 available students, 100 who met the eligibility criteria were selected to participate.

After obtaining informed consent, the students were randomly divided into the experimental and control groups. A simple randomization technique was used: numbered cards (1 to 100) were placed in a glass container, and the numbers were drawn and assigned alternately to the two groups. This method ensured equal allocation and reduced selection bias.

Based on the findings of a similar study and the mean comparison formula, with a Type I error of 0.05 and a power of 80%, the required sample size was 48 per group. To account for a potential 5% dropout rate, 50 participants were included in each group.

To minimize bias, a double-blind design was employed. The researcher who collected the data was unaware of group assignments. Similarly, the statistician who analyzed the data was blinded to the group allocations and treated the data as variables x₁ and x₂.

Tools of Data Collection:

To address the research objectives, data were collected using the following tools:

A) Demographic questionnaire:

Collected background information including age, gender, marital status, and academic history.

B) State-Trait Anxiety Inventory (STAI):

A 40-item self-report tool measuring both state and trait anxiety, with 20 items in each subscale. Items were scored on a 4-point Likert scale. Higher scores indicated greater anxiety. The STAI has demonstrated high validity and reliability in student populations.

C) Pre- and post-intervention anxiety scoring sheet:

Completed by students in both groups one week and two hours before their final exam.

Intervention:

Experimental Group:

Participants received both theoretical and practical training in Twin Heart Meditation from a certified researcher. They practiced meditation for 30 minutes per session, at least three times over a one-week period. Sessions were guided using MP3 audio recordings and conducted under the supervision of the researcher.

The intervention included:

Physical warm-up exercises (5 minutes) Heart chakra activation Crown chakra activation Blessing the Earth with loving-kindness Silent concentration on "Amen" Gratitude expression Closing exercises (5 minutes)

Control Group:

Participants received routine academic preparation without any additional intervention.

Implementation Phase:

The study was conducted in the Nursing Department of Near East University. After explaining the study procedures, written informed consent was obtained from all participants. Students were randomly assigned to either the intervention or control group. Meditation sessions were held in a quiet room. All participants completed the STAI questionnaire before and after the intervention period.

Ethical Considerations:

The study received approval from the Near East University Ethics Review Board under the approval number NUE/2023/114-1736. It adhered to the principles of the Declaration of Helsinki (1964). Participants were informed of their right to withdraw at any time without penalty. All participants provided written informed consent. Data confidentiality was strictly maintained throughout the study.

Statistical Analysis:

All data are analyzed using SPSS version 26. Descriptive statistics (mean, standard deviation, and frequencies) are used to summarize the data. Inferential statistical methods include:

Kolmogorov-Smirnov test to assess normality Paired t-test to evaluate pre- and post-intervention changes within each group Independent t-test to compare differences between the two groups Chi-square test or Fisher's exact test for analysis of categorical variables A significance level of P < 0.05 is considered statistically significant for all analyses.

ELIGIBILITY:
Inclusion criteria:

1. All seventh-semester undergraduate nursing students, both female and male, enrolled in the English-language program at the Department of Nursing, Near East University.
2. Students not using any other stress reduction methods, such as progressive muscle relaxation, pharmacological therapy, or similar techniques, to manage exam-related anxiety.
3. Students who voluntarily agreed to participate in the study and provided informed consent.

Exclusion criteria:

1. Doing meditation less than 3 times a week
2. Unwilling to continue cooperation in the project,
3. Using any psycho medicines (anti-depressants ...), mental health
4. Mourning, especially the death of loved ones or relatives in the 1st phase.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Test Anxiety Levels | Anxiety levels are measured at two time points-one week before the final exam and two hours before the final exam
  The primary outcome measure evaluates changes in exam-related anxiety levels among nursing students. Anxiety is measured using the State-Trait Anxiety Inventory (STAI), a validated psychological tool that assesses both temporary (state) and long-standing (trait) anxiety. The STAI includes two subscales, each with 20 items scored on a 4-point Likert scale. Higher scores indicate higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Pouran Varvani Farahani, PhD, Principal Investigator — PhD in Pediatric Nursing, Department of Nursing, Faculty of Health Science, Cyprus International University
Locations (1):
- Near East University, Nicosia, KKTC (Turkish Republic of Northern Cyprus),, Cyprus

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers